CLINICAL TRIAL: NCT07235605
Title: Intravenous Sedation and Analgesia Versus Local Anesthesia During Microwave Ablation of Benign Thyroid Nodules
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez University (Other)
Responsible Party: Principal Investigator, Ahmad Mohamed Ehab Moawd, Lecturer of Anesthesia, Intensive care, and pain medicine, Suez University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC.4.9.2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Benign Thyroid Nodule

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate to deep sedation (Experimental)
  Interventions: Procedure: Moderate to deep sedation
- Perithyroidal local anesthesia (Experimental)
  Interventions: Procedure: Perithyroidal local anesthesia

INTERVENTIONS:
Procedure: Moderate to deep sedation — Patients will receive drugs resulting in moderate to deep sedation, tailored to the specific portions of the procedure, which may offer potential benefits. This approach could provide patients with a potentially painless experience by utilizing moderate sedation during needle placement and deep sedation during the ablation phase. Additionally, this combination approach may minimize the risk of respiratory depression (which can be associated with TIVA and deep sedation) while promoting rapid recovery. The patients will receive premedication with the alpha-2-agonists, dexmedetomidine (2.5 μg/kg IV).
  Our combination approach will involve the use of fentanyl (1 microgram/kg), ketamine (1 milligram/ kg followed by 0.5 milligram/kg if repeated doses are necessary to accomplish longer duration) and propofol (Loading dose: 0.5-1 mg/kg, followed by top up doses of 30 mg to achieve deeper level of sedation or if the patient showed discomfort) to achieve sedation.
  Arms: Moderate to deep sedation
Procedure: Perithyroidal local anesthesia — the patients will be anesthetized by the physician performing ablation. After routine disinfection and draping, 10 ml of 1% lidocaine will be injected into the skin puncture site and thyroid capsule trans-mid-neck under US guidance. If the patient suffered from severe pain, 2-5ml of 1% lidocaine will be supplemented locally.
  Ablation will be discontinued when patients experienced unbearable pain
  Arms: Perithyroidal local anesthesia

SUMMARY:
The participants will be randomized into 2 equal groups by a computer-generated random numbers table, named group A and B. An independent data manager of computer-generated software will be responsible for randomization, assigning the participants to the groups using sequentially numbered, sealed, opaque envelopes containing computer-generated random numbers, accessible only to the anesthesiologist. The subjects will be randomly allocated to one of the two groups.

Group A: The participants will receive moderate to deep sedation.

Group B: The participants will receive perithyroidal local anesthesia.

History taking, clinical examination, and routine laboratory investigation will be performed preoperatively, and the participants will be instructed to fast for 6 hours preoperatively for solids and 2 hours for clear fluids. On arrival at the operation room, intravenous access will be established. ECG, noninvasive blood pressure, and arterial oxygen saturation will be monitored routinely. The Numerical Rating Scale (NRS) will be used to assess pain intensity. Preoperatively, all study subjects will be trained to use NRS pain scores.

In the intervention radiology room, a peripheral 20 G intravenous (IV) cannula will be inserted. The baseline parameters of five lead electrocardiogram (ECG), noninvasive blood pressure, and peripheral oxygen saturation will be recorded. A nasal oxygen cannula will be applied with a flow of 3 L/min.

In group A, participants will receive drugs resulting in moderate to deep sedation, tailored to the specific portions of the procedure, which may offer potential benefits. This approach could provide participants with a potentially painless experience by utilizing moderate sedation during needle placement and deep sedation during the ablation phase. Additionally, this combination approach may minimize the risk of respiratory depression (which can be associated with TIVA and deep sedation) while promoting rapid recovery. The participants will receive premedication with the alpha-2-agonists, dexmedetomidine (2.5 μg/kg IV).

The sedation combination approach will involve the use of fentanyl (1 microgram/kg), ketamine (1 milligram/ kg followed by 0.5 milligram/kg if repeated doses are necessary to accomplish longer duration) and propofol (Loading dose: 0.5-1 mg/kg, followed by top up doses of 30 mg to achieve deeper level of sedation or if the participant showed discomfort) to achieve sedation.

Deep sedation is defined as depression of the patient's consciousness such that they cannot be easily aroused but are able to respond purposefully following repeated or painful stimulation. Patients under deep sedation may have impaired ventilatory function and may require assistance maintaining a patent airway while Moderate sedation, defined as depressing the patient's consciousness while maintaining the ability to respond to verbal and tactile stimuli, is considered safe for various interventional radiology procedures. Patients under moderate sedation can maintain spontaneous respiration and a patent airway without assistance

Participants will be allowed to breathe spontaneously, and the propofol infusion rate will be titrated according to clinical response. Adequate sedation will be reached by the absence of body movements and failure to respond to verbal commands. Although participants cannot comply with breathing instructions. An oropharyngeal airway will be applied to avoid airway obstruction.

In group B, the participants will be anesthetized by the physician performing ablation. After routine disinfection and draping, 10 ml of 1% lidocaine will be injected into the skin puncture site and thyroid capsule trans-mid-neck under US guidance. If the participant suffered from severe pain, 2-5 ml of 1% lidocaine will be supplemented locally.

Ablation will be discontinued if participants experience unbearable pain.

All procedures will be performed by a single interventional radiologist (MD). Anesthesia will be administered by a single anesthesiologist (MD). Following asepsis protocols, the patients will undergo a procedure in which a linear ultrasound probe (10-15 MHz) LOGIQ P9 ultrasonography will be used. Microwave ablation will be done by Canyon Medical-Thyroid Ablation device.

Moving shot or fixed-applicator technique will be used based on the tumor characteristics. The target for ablation for a benign nodule will be the entire nodule. Nodules that are completely solid or mixed with 90% solid components will be directly ablated. For the solid nodules containing 50-89% of solid components, the cystic portion will be aspirated using a 20-23-G puncture needle before the ablation. For nodules with > 50% fluid content, the fluid will be withdrawn first, followed by saline flushing and ablation. The ablation procedure will be terminated when the target lesion is completely ablated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 60 years
* Both sexes
* American Society of Anesthesiologists (ASA)I-II.

Exclusion Criteria:

* Patients with chronic pain
* long-term alcoholism or taking tranquilizers or antipsychotic drugs
* Patients with malignant thyroid nodules
* Thyroid nodules compressing the trachea
* Hypertension in which BP was not controlled below 140/90 mmHg
* Patients with reflux esophagitis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
post-procedural pain 30 minutes after recovery by Numerical Rating Scale (NRS), and the pain level will be scored from 0 to 10, with 0 being the absence of pain and 10 being the worst pain. | 30 minutes after recovery from the procedure
  The primary objective of this study is to assess the post-procedural pain 30 minutes after recovery by the internationally accepted Numerical Rating Scale (NRS), and the pain level will be scored from 0 to 10, with 0 being the absence of pain and 10 being the worst pain.